CLINICAL TRIAL: NCT04659109
Title: A Randomized, Double Blind, Multicenter, Placebo Controlled, Parallel Group, Exploratory Efficacy and Safety Study of Glenzocimab in SARS-Cov-2-related Acute Respiratory Distress Syndrome
Brief Title: Glenzocimab in SARS-Cov-2 Acute Respiratory DistrEss syNdrome Related to COVID-19
Acronym: GARDEN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acticor Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACT-CS-006; 2020-002733-15 (EudraCT Number)
Record Dates: First submitted 2020-11-30; First posted 2020-12-09 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: SARS-CoV Infection; Acute Respiratory Distress Syndrome; COVID-19; ARDS
Keywords: Covid 19; ARDS; SARS-Cov; glenzocimab; Acute Respiratory Distress Syndrome; ACT017; glycoprotein VI; antiplatelet agent
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; Respiratory Distress Syndrome; COVID-19 | interventions — glenzocimab

STUDY DESIGN:
Intervention Model Description: A randomized, double blind, multicenter, placebo-controlled, parallel group, fixed dose, phase II study. The study evaluates the efficacy and safety of glenzocimab.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- glenzocimab 1000 mg (Experimental)
  Interventions: Drug: glenzocimab
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: glenzocimab — IV administration as a sterile product
  Other Names: ACT017
  Arms: glenzocimab 1000 mg
Drug: Placebo — IV administration
  Arms: Placebo

SUMMARY:
A randomized, double blind, multicenter, placebo-controlled, parallel group, fixed dose, phase II study to evaluate the efficacy and safety of glenzocimab in ARDS.

DETAILED DESCRIPTION:
This randomized, double blind, multicenter, placebo-controlled, parallel group, fixed dose, phase II study evaluates the efficacy and safety of glenzocimab in ARDS.

Patients will be screened for eligibility and all tests should have results prior to any randomization, so as to avoid screening failures to a maximum extent. The turn-around time for these tests should be comprised within 24hrs to allow for rapid inclusions if needed. Eligible patients (n=68) will be randomized in a 1:1 ratio to glenzocimab or placebo. Patient inclusions will be fractioned into sequential (3-day apart) cohorts of growing size (2, 4 then 6 patients), each balanced between glenzocimab and placebo in order to check safety in a gradual manner. A Data Safety Monitoring Board (DSMB) will meet after 12 patients will have been accrued, and again after the first 30 patients.

Glenzocimab will be administered by IV infusion. The dosing regimen will be 1000mg for 3 days. All patients will receive in parallel the best medical care at the discretion of the investigating center, or per local guidelines. The allocation of each patient in any given center to an active treatment or placebo will strictly follow a central randomization scheme. The study period will be of a maximum of 40 days per patient. Patients will be closely monitored during the first 7 days following randomization with complete evaluations being performed at 24 hrs, 48 hrs, 72 hrs, then on Days 4 (96 hrs), 5 (120 hrs), 7 (+/-1 day), 14 (+/-2 days), 20 (+/-2 days), 40 (+/-3 days). Should a patient being discharged before Day 40, distant consultations by telemedicine may be undertaken if it is not deemed desirable that the patient comes back to the institution.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female hospitalized patients ≥ 18 years (i.e., at least 18 years old at the time of randomization), having given their written consent.
2. Having a positive RT-PCR test for COVID-19
3. Presenting with symptoms of COVID-19, including:

   * Cough OR
   * Shortness of breath or difficulty breathing OR at least 2 of the following
   * Fever, defined as any body temperature 38°C
   * Chills
   * Repeated shaking with chills
   * Muscle pain
   * Headache
   * Sore throat
   * New loss of taste or smell
4. Presenting with signs of moderate but progressive pulmonary disease with:

   * respiratory symptoms (cough, dyspnea, etc.),
   * uni- or bilateral ground-glass opacities, or pulmonary infiltrates on chest radiograph and/or CT scan,
   * clinical and biological evidence of progression over the past 48hrs.
5. Effective birth control that should have been in place for at least 2 months in non-menopausal women and 4 months for men after IMP administration. Birth control methods considered to be highly effective include:

   * combined (estrogen-progestogen) hormonal contraception associated with the inhibition of ovulation: oral, intravaginal, transdermal,
   * progesterone-only hormonal contraception associated with the inhibition of ovulation: oral, injectable, implantable,
   * intrauterine device,
   * intrauterine hormone-releasing system,
   * bilateral tubal occlusion,
   * vasectomized partner.
6. Women of child-bearing potential must have negative results of a urinary or plasma pregnancy test (serum HCG).

Exclusion Criteria:

1. Patients requiring immediate admission to the ICU,
2. Patients requiring invasive mechanical ventilation,
3. ARDS of another origin,
4. Concomitant pulmonary infection (pneumoniae) with another agent, notably bacterial or fungal,
5. Patients under immunosuppressive agents,
6. Childbirth within <10 days,
7. Pregnancy or breastfeeding,
8. Prior cardiopulmonary resuscitation <10 days,
9. Allergy or hypersensitivity to drugs of the same class
10. Participation in another interventional clinical trial within 30 days prior to the inclusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2021-08-06 (Actual); Study Completion 2021-08-06 (Actual)

PRIMARY OUTCOMES:
Progression from moderate to severe respiratory distress assessed at Day 4 | Day 4
  Progression from moderate to severe assessed at Day 4 is a composite failure endpoint defined as the occurrence of at least one of the following failure events :
  * Respiratory rate (RR) ≥ 30/min, or
  * Oxygen Saturation (SpO2) ≤ 93% in resting state, or
  * Oxygen Pressure/ Inspired fraction (PaO2/FiO2) ≤ 200mmHg
  * Death occurring prior to or on Day 4

SECONDARY OUTCOMES:
All cause mortality at day 40 | Day 40 (maximum)
WHO-COVID-19 Scale | Up to Day 40
  WHO COVID-19 Ordinal Scoring Scale is 9 point ordinal scale
NEWS-2 Scale | Up to Day 40
  Determines the degree of illness of a patient and prompts critical care intervention (recommended by NHS over original NEWS): total possible score ranges from 0 to 20. The higher the scores the greater the clinical risk.
Respiratory Rate status (RR) | Up to Day 40
  Respiratory Rate status defined as:: o Normal:<20/min,
  * Mild:20/min≤RR<24/min,
  * Moderate:24/min≤RR<30/min, o Severe:≥30/min,
  * Death.
Hypoxemia status | Up to Day 40
  Hypoxemia status defined as:: o Normal:>300mmHg,
  * Mild: 200 mmHg < PaO2/FiO2 ≤ 300 mmHg,
  * Moderate:100mmHg<PaO2/FIO2≤200mmHg, o Severe:PaO2/FIO2≤100mmHg,
  * Death.
SpO2 status | Up to Day 40
  SpO2 status defined as: o Normal:>95%
  * Mild:93%<SpO2≤95%,
  * Moderate:90%<SpO2≤93%, o Severe:≤90%,
  * Death.
CHEST CT-Scan (or in exceptional cases, chest radiogram) | Day 4
Oxygen-free days | Up to Day 40
Admission to the ICU | Up to Day 40
ICU-free days | Up to Day 40
Hospital-free days | Up to Day 40
Clinical recovery and Time to Clinical recovery | Up to Day 40
Cure and Time-to-cure | Up to Day 40
Incidence, nature and severity of Adverse Events, SAEs, SUSARs and Treatment-Emergent Adverse Events (TEAEs) | Up to Day 40
Incidence of bleeding-related events | Up to Day 40
Incidence of hypersensitivity reactions | Up to Day 40
Changes from baseline on blood pressure | Up to Day 40
Changes from baseline on heart rate | Up to Day 40
Changes from baseline on NFS | Up to Day 40
Changes from baseline on INR/PTT | Up to Day 40
Changes from baseline on platelet count | Up to Day 40
Changes from baseline on plasma fibrinogen level | Up to Day 40
Changes from baseline on plasma D-Dimers level | Up to Day 40
Changes from baseline on serum-glucose level | Up to Day 40
Changes from baseline on urea level | Up to Day 40
Changes from baseline on creatinemia | Up to Day 40
Changes from baseline on LFTs (ASAT/ALAT) | Up to Day 40
Changes from baseline on CRP level | Up to Day 40
Changes from baseline on LDH level | Up to Day 40
Changes from baseline on IL6 level | Up to Day 40
Changes from baseline on Tnt | Up to Day 40
Changes from baseline on NT proBNP | Up to Day 40
Changes from baseline on procalcitonin level | Up to Day 40
Changes from baseline on ferritin level | Up to Day 40
ECG over the course of the study versus screening | Up to Day 40
  Changes in one or several of the usual ECG parameters compared to baseline or screening, i.e. sinusal rhythm, cardiac axis, QRS value, QT/QTc segment, Wave direction, and any abnormality.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital de Hautepierre, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Renaud L, Lebozec K, Voors-Pette C, Dogterom P, Billiald P, Jandrot Perrus M, Pletan Y, Machacek M. Population Pharmacokinetic/Pharmacodynamic Modeling of Glenzocimab (ACT017) a Glycoprotein VI Inhibitor of Collagen-Induced Platelet Aggregation. J Clin Pharmacol. 2020 Sep;60(9):1198-1208. doi: 10.1002/jcph.1616. Epub 2020 Jun 4. PMID 32500636
- [Background] Voors-Pette C, Lebozec K, Dogterom P, Jullien L, Billiald P, Ferlan P, Renaud L, Favre-Bulle O, Avenard G, Machacek M, Pletan Y, Jandrot-Perrus M. Safety and Tolerability, Pharmacokinetics, and Pharmacodynamics of ACT017, an Antiplatelet GPVI (Glycoprotein VI) Fab. Arterioscler Thromb Vasc Biol. 2019 May;39(5):956-964. doi: 10.1161/ATVBAHA.118.312314. PMID 31017822